CLINICAL TRIAL: NCT03321565
Title: Johns Hopkins Weight Management Center Patient Data
Acronym: JHWMC
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: JH WMC patient data
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Behavioral counseling and optional meal replacement program — Medical assessment and medical supervision of weight loss Measurements of metabolism and body composition Individualized exercise programs Personal training Support group meetings Individual psychotherapy A variety of nutritional plans including meal replacement options Nutrition education Long-term weight maintenance and relapse prevention programs

SUMMARY:
Patient records from Johns Hopkins Weight Management Center historical files

DETAILED DESCRIPTION:
Examination of historical patient files from the Johns Hopkins Weight Management Center, to be conducted by a study team led by the attending physician and director of the Center. Analyses will examine weight-related outcomes based on participation in the Weight Management Center program.

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a patient at the Johns Hopkins Weight Management Center

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who enroll themselves at the Johns Hopkins Weight Management Center, with the goal of reaching or maintaining a healthy BMI.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1990-2020
  Weight-related measures for patients of the Johns Hopkins Weight Management Center.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Weight Management Center, Baltimore, Maryland, United States